CLINICAL TRIAL: NCT01156142
Title: A Randomized Double-Blind Study of Doxepin Rinse Versus Placebo in the Treatment of Acute Oral Mucositis Pain in Patients Receiving Radiotherapy With or Without Chemotherapy
Brief Title: Doxepin Hydrochloride in Treating Oral Mucositis Pain in Patients With Head and Neck Cancer Undergoing Radiation Therapy With or Without Chemotherapy
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Alliance for Clinical Trials in Oncology (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Supportive Care
Other Study IDs: NCCTG-N09C6; NCI-2011-02049 (Registry Identifier: CTRP (Clinical Trials Reporting System)); CDR0000675520 (Registry Identifier: PDQ (Physician Data Query)); U10CA037404 (NIH)
Record Dates: First submitted 2010-07-01; First posted 2010-07-02 (Estimated); Results first posted 2017-05-08 (Actual); Last update posted 2017-08-09 (Actual); Status verified 2017-07

CONDITIONS: Head and Neck Cancer; Mucositis; Oral Complications of Radiation Therapy; Pain
Keywords: oral complications of radiation therapy; mucositis; pain; stage I squamous cell carcinoma of the paranasal sinus and nasal cavity; recurrent squamous cell carcinoma of the hypopharynx; squamous cell carcinoma of the hypopharynx; recurrent squamous cell carcinoma of the larynx; recurrent verrucous carcinoma of the larynx; squamous cell carcinoma of the larynx; verrucous carcinoma of the larynx; recurrent adenoid cystic carcinoma of the oral cavity; recurrent mucoepidermoid carcinoma of the oral cavity; recurrent verrucous carcinoma of the oral cavity; adenoid cystic carcinoma of the oral cavity; mucoepidermoid carcinoma of the oral cavity; verrucous carcinoma of the oral cavity; squamous cell carcinoma of the lip and oral cavity; recurrent basal cell carcinoma of the lip; recurrent squamous cell carcinoma of the lip and oral cavity; basal cell carcinoma of the lip; metastatic squamous neck cancer with occult primary squamous cell carcinoma; recurrent metastatic squamous neck cancer with occult primary; untreated metastatic squamous neck cancer with occult primary; recurrent lymphoepithelioma of the nasopharynx; recurrent squamous cell carcinoma of the nasopharynx; lymphoepithelioma of the nasopharynx; squamous cell carcinoma of the nasopharynx; recurrent lymphoepithelioma of the oropharynx; recurrent squamous cell carcinoma of the oropharynx; lymphoepithelioma of the oropharynx; squamous cell carcinoma of the oropharynx; recurrent esthesioneuroblastoma of the paranasal sinus and nasal cavity; recurrent inverted papilloma of the paranasal sinus and nasal cavity; recurrent midline lethal granuloma of the paranasal sinus and nasal cavity; recurrent squamous cell carcinoma of the paranasal sinus and nasal cavity; esthesioneuroblastoma of the paranasal sinus and nasal cavity; inverted papilloma of the paranasal sinus and nasal cavity; midline lethal granuloma of the paranasal sinus and nasal cavity; squamous cell carcinoma of the paranasal sinus and nasal cavity; high-grade salivary gland mucoepidermoid carcinoma; low-grade salivary gland mucoepidermoid carcinoma; recurrent salivary gland cancer; salivary gland acinic cell tumor; salivary gland adenocarcinoma; salivary gland adenoid cystic carcinoma; salivary gland anaplastic carcinoma; salivary gland malignant mixed cell type tumor; salivary gland poorly differentiated carcinoma; salivary gland squamous cell carcinoma; salivary gland cancer; tongue cancer
MeSH Terms: conditions — Head and Neck Neoplasms; Mucositis; Pain; Squamous Cell Carcinoma of Head and Neck; Esthesioneuroblastoma, Olfactory; Salivary Gland Neoplasms; Tongue Neoplasms | interventions — Doxepin

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Arm I (Experimental): Patients receive doxepin hydrochloride oral rinse (swish, gargle, and spit) over 1 minute on day 1. Patients may crossover to arm II on day 2.
  Interventions: Drug: doxepin hydrochloride
- Arm II (Placebo Comparator): Patients receive placebo oral rinse (swish, gargle, and spit) over 1 minute on day 1. Patients may crossover to arm I on day 2.
  Interventions: Other: placebo

INTERVENTIONS:
Drug: doxepin hydrochloride — Oral rinse
  Arms: Arm I
Other: placebo — Oral rinse
  Arms: Arm II

SUMMARY:
RATIONALE: Doxepin hydrochloride may be an effective treatment for oral mucositis pain in patients undergoing radiation therapy with or without chemotherapy.

PURPOSE: This randomized phase III trial is studying doxepin hydrochloride to see how well it works compared to placebo in treating oral mucositis pain in patients with head and neck cancer undergoing radiation therapy with or without chemotherapy.

DETAILED DESCRIPTION:
OUTLINE: This is a multicenter study. Patients are stratified according to gender, concurrent radiosensitizing chemotherapy (yes vs no), and age (< 60 years vs ≥ 60 years). Patients are randomized to 1 of 2 treatment arms.

* Arm I: Patients receive doxepin hydrochloride oral rinse (swish, gargle, and spit)* over 1 minute on day 1. Patients may crossover to arm II on day 2.
* Arm II: Patients receive placebo oral rinse (swish, gargle, and spit)* over 1 minute on day 1.

Patients may crossover to arm I on day 2. The primary and secondary objectives are detailed below.

Primary Objective:

Determine whether doxepin oral rinse is effective in reducing OM-related pain in patients undergoing RT to the oral cavity, as measured by a patient-reported questionnaire at 5,15, 30, 60, 120 and 240 minutes

Secondary Objectives:

1. Assess the adverse event profile of doxepin rinse using a patient-reported questionnaire at 5, 15, 30, 60, 120 and 240 minutes for domains of unpleasant taste, burning or stinging discomfort, and drowsiness.
2. Compare the incidence of using alternative analgesics before 4 hours, between the doxepin oral rinse and placebo arms.
3. Assess patient preference for continued therapy with oral rinse after initial test rinse or after the cross-over phase.

NOTE: * Patients are instructed to avoid taking medications for mucositis pain 60 minutes before and after study medication.

After completing study therapy, patients have the option to receive doxepin hydrochloride oral rinse every 4 hours as needed during radiotherapy.

Patients complete questionnaires at baseline, and at 5, 15, 30, 60, 120, and 240 minutes after study medication. Patients who choose to continue doxepin hydrochloride oral rinse also complete weekly questionnaires.

ELIGIBILITY:
Inclusion Criteria:

1. ≥ 18 years of age
2. Histologic proof of malignancy currently undergoing a course of RT (with or without chemotherapy) to a dose of ≥ 5000 cGy using 1.60 to 2.20 Gy per fraction. Note: At least one third of the oral cavity mucosa must be included in the radiation therapy fields.
3. ≥ 4 oral pain felt to be related to mucositis for which the patient wants relief as measured by the Numeric Measure of Oral Pain. Note: An oral exam confirming the presence of mucositis should be performed by the enrolling clinician in addition to patient feedback.
4. Ability to complete questionnaire(s) independently or with assistance
5. ECOG Performance Status 0, 1 or 2.
6. Provide informed written consent.
7. Willingness to return to enrolling institution for follow-up.

Exclusion Criteria:

1. Known allergy to doxepin, tricyclic antidepressants, or any known component of the drug formulation
2. Use of a tricyclic antidepressant or monoamine oxidase inhibitor within the 2 weeks prior to registration
3. Current untreated or unresolved oral candidiasis or oral HSV infection
4. Current untreated narrow angle glaucoma
5. Current untreated urinary retention ≤ 6 weeks prior to registration
6. Co-morbid systemic illnesses or other severe concurrent disease which, in the judgment of the investigator, would make the patient inappropriate for entry into this study or interfere significantly with the proper assessment of safety and toxicity of the prescribed regimens
7. Any of the following because this study involves a study agent whose genotoxic, mutagenic and teratogenic effects on the developing fetus and newborn are unknown:

   * Pregnant women
   * Nursing women
   * Men or women of childbearing potential who are unwilling to employ adequate contraception

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 155 (Actual)
Dates: Start 2010-12; Primary Completion 2012-05 (Actual); Study Completion 2015-03-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Robert C. Miller, MD, Study Chair — Mayo Clinic
Locations (120):
- United States (120):
  - Mayo Clinic Scottsdale, Scottsdale, Arizona
  - Saint Francis/Mount Sinai Regional Cancer Center at Saint Francis Hospital and Medical Center, Hartford, Connecticut
  - Mayo Clinic - Jacksonville, Jacksonville, Florida
  - MBCCOP - Medical College of Georgia Cancer Center, Augusta, Georgia
  - Saint Alphonsus Cancer Care Center at Saint Alphonsus Regional Medical Center, Boise, Idaho
  - CCOP - Carle Cancer Center, Urbana, Illinois
  - Elkhart Clinic, LLC, Elkhart, Indiana
  - Michiana Hematology-Oncology, PC - Elkhart, Elkhart, Indiana
  - Elkhart General Hospital, Elkhart, Indiana
  - Howard Community Hospital, Kokomo, Indiana
  - Center for Cancer Therapy at LaPorte Hospital and Health Services, La Porte, Indiana
  - Indiana University Health La Porte Hospital, La Porte, Indiana
  - Michiana Hematology-Oncology, PC - South Bend, Mishawaka, Indiana
  - Saint Joseph Regional Medical Center, Mishawaka, Indiana
  - Michiana Hematology Oncology PC-Mishawaka, Mishawaka, Indiana
  - Michiana Hematology Oncology PC - Plymouth, Plymouth, Indiana
  - CCOP - Northern Indiana CR Consortium, South Bend, Indiana
  - Memorial Hospital of South Bend, South Bend, Indiana
  - Michiana Hematology Oncology PC - La Porte, Westville, Indiana
  - McFarland Clinic, PC, Ames, Iowa
  - Cedar Rapids Oncology Associates, Cedar Rapids, Iowa
  - Mercy Regional Cancer Center at Mercy Medical Center, Cedar Rapids, Iowa
  - Boston University Cancer Research Center, Boston, Massachusetts
  - Hickman Cancer Center at Bixby Medical Center, Adrian, Michigan
  - Saint Joseph Mercy Cancer Center, Ann Arbor, Michigan
  - CCOP - Michigan Cancer Research Consortium, Ann Arbor, Michigan
  - Battle Creek Health System Cancer Care Center, Battle Creek, Michigan
  - Mecosta County Medical Center, Big Rapids, Michigan
  - Oakwood Cancer Center at Oakwood Hospital and Medical Center, Dearborn, Michigan
  - Saint John Hospital and Medical Center, Detroit, Michigan
  - Genesys Hurley Cancer Institute, Flint, Michigan
  - Hurley Medical Center, Flint, Michigan
  - Genesys Regional Medical Center, Grand Blanc, Michigan
  - Butterworth Hospital at Spectrum Health, Grand Rapids, Michigan
  - CCOP - Grand Rapids, Grand Rapids, Michigan
  - Lacks Cancer Center at Saint Mary's Health Care, Grand Rapids, Michigan
  - Van Elslander Cancer Center at St. John Hospital and Medical Center, Grosse Pointe Woods, Michigan
  - Allegiance Health, Jackson, Michigan
  - Foote Memorial Hospital, Jackson, Michigan
  - Sparrow Regional Cancer Center, Lansing, Michigan
  - St. Mary Mercy Hospital, Livonia, Michigan
  - Community Cancer Center of Monroe, Monroe, Michigan
  - Mercy Memorial Hospital - Monroe, Monroe, Michigan
  - Mercy General Health Partners, Muskegon, Michigan
  - St. Joseph Mercy Oakland, Pontiac, Michigan
  - Mercy Regional Cancer Center at Mercy Hospital, Port Huron, Michigan
  - Seton Cancer Institute at Saint Mary's - Saginaw, Saginaw, Michigan
  - Lakeland Regional Cancer Care Center - St. Joseph, Saint Joseph, Michigan
  - Lakeside Cancer Specialists, PLLC, Saint Joseph, Michigan
  - Marie Yeager Cancer Center, Saint Joseph, Michigan
  - Munson Medical Center, Traverse City, Michigan
  - St. John Macomb Hospital, Warren, Michigan
  - MeritCare Bemidji, Bemidji, Minnesota
  - Sanford Clinic North-Bemidgi, Bemidji, Minnesota
  - Fairview Ridges Hospital, Burnsville, Minnesota
  - Mercy and Unity Cancer Center at Mercy Hospital, Coon Rapids, Minnesota
  - Fairview Southdale Hospital, Edina, Minnesota
  - Mercy and Unity Cancer Center at Unity Hospital, Fridley, Minnesota
  - Hutchinson Area Health Care, Hutchinson, Minnesota
  - HealthEast Cancer Care at St. John's Hospital, Maplewood, Minnesota
  - Minnesota Oncology - Maplewood, Maplewood, Minnesota
  - Virginia Piper Cancer Institute at Abbott - Northwestern Hospital, Minneapolis, Minnesota
  - Hennepin County Medical Center - Minneapolis, Minneapolis, Minnesota
  - New Ulm Medical Center, New Ulm, Minnesota
  - Humphrey Cancer Center at North Memorial Outpatient Center, Robbinsdale, Minnesota
  - Mayo Clinic Cancer Center, Rochester, Minnesota
  - CCOP - Metro-Minnesota, Saint Louis Park, Minnesota
  - Park Nicollet Cancer Center, Saint Louis Park, Minnesota
  - Regions Hospital Cancer Care Center, Saint Paul, Minnesota
  - United Hospital, Saint Paul, Minnesota
  - St. Francis Cancer Center at St. Francis Medical Center, Shakopee, Minnesota
  - Lakeview Hospital, Stillwater, Minnesota
  - Ridgeview Medical Center, Waconia, Minnesota
  - Willmar Cancer Center at Rice Memorial Hospital, Willmar, Minnesota
  - Minnesota Oncology - Woodbury, Woodbury, Minnesota
  - Cancer Resource Center - Lincoln, Lincoln, Nebraska
  - CCOP - Missouri Valley Cancer Consortium, Omaha, Nebraska
  - Immanuel Medical Center, Omaha, Nebraska
  - Alegant Health Cancer Center at Bergan Mercy Medical Center, Omaha, Nebraska
  - Lakeside Hospital, Omaha, Nebraska
  - Creighton University Medical Center, Omaha, Nebraska
  - MeritCare Broadway, Fargo, North Dakota
  - Sanford Clinic North-Fargo, Fargo, North Dakota
  - CCOP - MeritCare Hospital, Fargo, North Dakota
  - Roger Maris Cancer Center at MeritCare Hospital, Fargo, North Dakota
  - Sanford Medical Center-Fargo, Fargo, North Dakota
  - Altru Cancer Center at Altru Hospital, Grand Forks, North Dakota
  - Wood County Oncology Center, Bowling Green, Ohio
  - Community Cancer Center, Elyria, Ohio
  - Hematology Oncology Center, Elyria, Ohio
  - Lima Memorial Hospital, Lima, Ohio
  - Northwest Ohio Oncology Center, Maumee, Ohio
  - St. Charles Mercy Hospital, Oregon, Ohio
  - Toledo Clinic - Oregon, Oregon, Ohio
  - Flower Hospital Cancer Center, Sylvania, Ohio
  - Mercy Hospital of Tiffin, Tiffin, Ohio
  - Toledo Hospital, Toledo, Ohio
  - St. Vincent Mercy Medical Center, Toledo, Ohio
  - Medical University of Ohio Cancer Center, Toledo, Ohio
  - CCOP - Toledo Community Hospital, Toledo, Ohio
  - St. Anne Mercy Hospital, Toledo, Ohio
  - Toledo Clinic, Incorporated - Main Clinic, Toledo, Ohio
  - Fulton County Health Center, Wauseon, Ohio
  - Fredericksburg Oncology, Incorporated, Fredericksburg, Virginia
  - Marshfield Clinic - Chippewa Center, Chippewa Falls, Wisconsin
  - Center for Cancer Treatment & Prevention at Sacred Heart Hospital, Eau Claire, Wisconsin
  - Marshfield Clinic Cancer Care at Regional Cancer Center, Eau Claire, Wisconsin
  - Marshfield Clinic - Ladysmith Center, Ladysmith, Wisconsin
  - Marshfield Clinic - Marshfield Center, Marshfield, Wisconsin
  - Saint Joseph's Hospital, Marshfield, Wisconsin
  - Marshfield Clinic - Lakeland Center, Minocqua, Wisconsin
  - Ministry Medical Group at Saint Mary's Hospital, Rhinelander, Wisconsin
  - Marshfield Clinic - Indianhead Center, Rice Lake, Wisconsin
  - Marshfield Clinic at Saint Michael's Hospital, Stevens Point, Wisconsin
  - Saint Michael's Hospital Cancer Center, Stevens Point, Wisconsin
  - Marshfield Clinic - Wausau Center, Wausau, Wisconsin
  - Diagnostic and Treatment Center, Weston, Wisconsin
  - Marshfield Clinic - Weston Center, Weston, Wisconsin
  - Ministry Saint Clare's Hospital, Weston, Wisconsin
  - Marshfield Clinic - Wisconsin Rapids Center, Wisconsin Rapids, Wisconsin

REFERENCES:
- [Derived] Leenstra JL, Miller RC, Qin R, Martenson JA, Dornfeld KJ, Bearden JD, Puri DR, Stella PJ, Mazurczak MA, Klish MD, Novotny PJ, Foote RL, Loprinzi CL. Doxepin rinse versus placebo in the treatment of acute oral mucositis pain in patients receiving head and neck radiotherapy with or without chemotherapy: a phase III, randomized, double-blind trial (NCCTG-N09C6 [Alliance]). J Clin Oncol. 2014 May 20;32(15):1571-7. doi: 10.1200/JCO.2013.53.2630. Epub 2014 Apr 14. PMID 24733799

RESULTS

PARTICIPANT FLOW:
Groups:
- Arm I (Doxepin-Placebo): Patients receive (10 mg/mL x 2.5 mL) 25 mg doxepin hydrochloride (diluted to 5 mL with 2.5 mL of sterile water for irrigation, or sterile water for injection, or distilled water) oral rinse (swish, gargle, and spit) over 1 minute on day 1. Patients may crossover to arm II on day 2.
- Arm II (Placebo-Doxepin): Patients receive 2.5 mL placebo (diluted to 5 mL with 2.5 mL of sterile water for irrigation, or sterile water for injection, or distilled water) oral rinse (swish, gargle, and spit) over 1 minute on day 1. Patients may crossover to arm I on day 2.
Period: Overall Study
Arm/Group | Arm I (Doxepin-Placebo) | Arm II (Placebo-Doxepin)
Started | 77 | 78
Completed | 69 | 71
Not Completed | 8 | 7
Not completed — Withdrawal by Subject | 8 | 6
Not completed — Ineligible | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Arm I (Doxepin-Placebo) | Arm II (Placebo-Doxepin) | Total
Number analyzed (Participants) | 69 | 71 | 140
Age, Continuous [Mean (Full Range); unit: years] | 62 [39.0 to 93.0] | 60 [37.0 to 86.0] | 61 [37.0 to 93.0]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 13 | 15 | 28
  Male | 56 | 56 | 112
Region of Enrollment [Number; unit: participants]
  United States | 69 | 71 | 140

OUTCOME MEASURES:

1. Primary Outcome: Total Pain Reduction (Mouth and Throat)
Description: The total pain reduction will be calculated by the (average of mouth and throat) area under the curve (AUC) adjusting for baseline, with time scale replaced by a numerical scale of 1,2,3,4,5,6. The numerical scale will be used rather than the raw time scale in order to give proper weights to more immediate patient-reported mouth pain outcomes after treatment. The AUC will be calculated by proration when there are terminal missing data. If the missing data are intermittent, simple imputation will be applied to calculate the AUC. The question ('On a scale from 0 to 10, what number best describes your MOUTH PAIN due to your radiation treatment now?') used 11-point numerical analog scales (0 (no pain) to 10 (worst pain imaginable or possible) scores) to measure pain. The AUCs for the two treatment arms were compared by using the Wilcoxon rank sum test with 95% CIs.
Time Frame: Baseline and Day 1
Population: If a patient cancels, is missing baseline data, or only provides baseline data, he/she will be excluded from the statistical analysis. The primary analysis of the total pain reduction will only use primary data from the first phase.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Arm I (Doxepin-Placebo) | Arm II (Placebo-Doxepin)
Number analyzed (Participants) | 69 | 71
units on a scale | -9.1 (7.9) | -4.7 (6.1)
Statistical Analysis 1: Comparison: Arm I (Doxepin-Placebo) vs Arm II (Placebo-Doxepin); Test type: Superiority or Other; p < 0.001, Wilcoxon (Mann-Whitney); Mean Difference (Final Values) = -4.4, 95% CI 2-sided [-6.7 to -2.1]

2. Secondary Outcome: Total Taste of the Oral Rinse
Description: The total taste of the oral rinse will be calculated by the area under the curve (AUC) adjusting for baseline, with time scale replaced by a numerical scale of 1,2,3,4,5,6 , and analyzed in the same way as the primary endpoint. The numerical scale will be used rather than the raw time scale in order to give proper weights to more immediate patient-reported mouth pain outcomes after treatment. The AUC will be calculated by proration when there are terminal missing data. If the missing data are intermittent, simple imputation will be applied to calculate the AUC. The question ('On a scale from 0 to 10, what number best describes the TASTE OF THE ORAL RINSE now?') used 11-point numerical analog scales (0 (acceptable taste) to 10(terrible taste), with higher values representing worse outcome) to evaluate the total taste of the oral rinse. The AUCs for the two treatment arms were compared by using the Wilcoxon rank sum test with 95% CIs.
Time Frame: Up to 9 days
Population: If a patient cancels, is missing baseline data, or only provides baseline data, he/she will be excluded from the statistical analysis.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Arm I (Doxepin-Placebo) | Arm II (Placebo-Doxepin)
Number analyzed (Participants) | 69 | 71
units on a scale | 7.7 (7.1) | 5.1 (7.7)
Statistical Analysis 1: Comparison: Arm I (Doxepin-Placebo) vs Arm II (Placebo-Doxepin); Test type: Superiority or Other; p = 0.0018, Wilcoxon (Mann-Whitney); Mean Difference (Final Values) = 2.6, 95% CI 2-sided [0.1 to 5.1]

3. Secondary Outcome: Total Stinging or Burning From the Oral Rinse
Description: The total stinging or burning from the oral rinse will be calculated by the area under the curve (AUC) adjusting for baseline, with time scale replaced by a numerical scale of 1,2,3,4,5,6. The numerical scale will be used rather than the raw time scale in order to give proper weights to more immediate patient-reported mouth pain outcomes after treatment. The AUC will be calculated by proration when there are terminal missing data. If the missing data are intermittent, simple imputation will be applied to calculate the AUC. The question ('On a scale from 0 to 10, what number best describes any STINGING OR BURNING FROM THE ORAL RINSE now?') used 11-point numerical analog scales (0 (no stinging or burning) to 10 (worst stinging or burning possible) scores) to total stinging or burning from the oral rinse. The AUCs for the two treatment arms were compared by using the Wilcoxon rank sum test with 95% CIs.The statistical analysis will be the same as the primary analysis.
Time Frame: Up to 9 days
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Arm I (Doxepin-Placebo) | Arm II (Placebo-Doxepin)
Number analyzed (Participants) | 69 | 71
units on a scale | 9.6 (8.4) | 4.0 (8.0)
Statistical Analysis 1: Comparison: Arm I (Doxepin-Placebo) vs Arm II (Placebo-Doxepin); Test type: Superiority or Other; p = 0.001, Wilcoxon (Mann-Whitney); Mean Difference (Final Values) = 5.6, 95% CI 2-sided [2.9 to 8.3]

4. Secondary Outcome: Total Drowsiness Increase
Description: The total drowsiness increase will be calculated by the area under the curve (AUC) adjusting for baseline, with time scale replaced by a numerical scale of 1,2,3,4,5,6. The numerical scale will be used rather than the raw time scale in order to give proper weights to more immediate patient-reported mouth pain outcomes after treatment. The AUC will be calculated by proration when there are terminal missing data. If the missing data are intermittent, simple imputation will be applied to calculate the AUC. The question ('On a scale from 0 to 10, what number best describes your DROWSINESS now?') used 11-point numerical analog scales (0 (no drowsiness) to 10 (extreme drowsiness, leading to sleep) scores) to measure total drowsiness increase. The AUCs for the two treatment arms were compared by using the Wilcoxon rank sum test with 95% CIs. The statistical analysis will be the same as the primary analysis.
Time Frame: Up to 9 days
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Arm I (Doxepin-Placebo) | Arm II (Placebo-Doxepin)
Number analyzed (Participants) | 69 | 71
units on a scale | -0.7 (10.3) | -2.4 (6.6)
Statistical Analysis 1: Comparison: Arm I (Doxepin-Placebo) vs Arm II (Placebo-Doxepin); Test type: Superiority or Other; p = 0.0297, Wilcoxon (Mann-Whitney); Mean Difference (Final Values) = 1.7, 95% CI 2-sided [-1.2 to 4.6]

5. Secondary Outcome: Incidence of Using Alternative Analgesics Between 2 and 4 Hours After the Initial Mouthwash
Description: The incidence of utilizing additional analgesics between 2 and 4 hours after the initial mouthwash will be compared between the arms by the Chi-square test .
Time Frame: Up to 9 days
Measure: Number; unit: percentage of patients
Arm/Group | Arm I (Doxepin-Placebo) | Arm II (Placebo-Doxepin)
Number analyzed (Participants) | 69 | 71
percentage of patients
  At 2 hours after the initial mouthwash | 8.8 | 2.9
  At 4 hours after the initial mouthwash | 16.9 | 14.5
Statistical Analysis 1: Comparison: Arm I (Doxepin-Placebo) vs Arm II (Placebo-Doxepin); At 2 hours after initial mouthwash; Test type: Superiority or Other; p = 0.1392, Chi-squared
Statistical Analysis 2: Comparison: Arm I (Doxepin-Placebo) vs Arm II (Placebo-Doxepin); At 4 hours after initial mouthwash; Test type: Superiority or Other; p = 0.6989, Chi-squared

6. Secondary Outcome: Patient Preference for Continuing Therapy With Oral Doxepin Hydrochloride
Description: After each dose was administered, patients were asked if they would like to continue rinses with that particular agent. The percentage of patients who expressed an interest in continuing therapy are reported below.
Time Frame: Up to 9 days
Measure: Number; unit: percentage of patients
Arm/Group | Arm I (Doxepin-Placebo) | Arm II (Placebo-Doxepin)
Number analyzed (Participants) | 69 | 71
percentage of patients | 77.3 | 51.5
Statistical Analysis 1: Comparison: Arm I (Doxepin-Placebo) vs Arm II (Placebo-Doxepin); Test type: Superiority or Other; p = 0.0018, Chi-squared

ADVERSE EVENTS:
Time Frame: Adverse events are assessed during the Active Monitoring Phase at the following time points: at time Dose 1 of study treatment is administered, at time of Dose 2 crossover, during the Optional Continuation Phase, and at the end of the study. All adverse events are collected during the first day; up to 9 days.
Description: The descriptions and grading scales found in the revised NCI Common Terminology Criteria for Adverse Events (CTCAE) version 4.0 will be utilized for AE reporting. All graded adverse events are reported.
Arm/Group | Arm I (Doxepin-Placebo) | Arm II (Placebo-Doxepin)
Serious Adverse Events (participants affected / at risk) | 0/74 | 0/75
Other Adverse Events (participants affected / at risk) | 10/74 | 8/75
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm I (Doxepin-Placebo) (N=74) | Arm II (Placebo-Doxepin) (N=75)
Diarrhea (Gastrointestinal disorders) | 1 (1) | 0 (0)
Dry mouth (Gastrointestinal disorders) | 3 (4) | 0 (0)
Dysphagia (Gastrointestinal disorders) | 1 (1) | 0 (0)
Mucositis oral (Gastrointestinal disorders) | 4 (9) | 6 (12)
Nausea (Gastrointestinal disorders) | 1 (1) | 1 (2)
Oral pain (Gastrointestinal disorders) | 2 (5) | 2 (2)
Salivary duct inflammation (Gastrointestinal disorders) | 1 (1) | 0 (0)
Vomiting (Gastrointestinal disorders) | 0 (0) | 1 (2)
Fatigue (General disorders) | 1 (1) | 0 (0)
Anorexia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 1 (2)
Lethargy (Nervous system disorders) | 0 (0) | 1 (1)
Somnolence (Nervous system disorders) | 1 (1) | 2 (2)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes